CLINICAL TRIAL: NCT02543840
Title: Hybrid Controlled Trial to Implement Collaborative Care in General Mental Health
Brief Title: Hybrid Collaborative Care Randomized Program Evaluation
Acronym: BHIP-CCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Bauer, Associate Director, Center for Healthcare Organization and Implementation Research, VA Boston Healthcare System
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-289; QUE-15-289 (Other: U.S. Department of Veterans Affairs)
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Mental Health Disorders
Keywords: Quality Improvement; Organization of Services; Implementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation Facilitation (Experimental): Implementation Facilitation consists of the Center for Disease Control's Replicating Effective Programs, plus External Facilitation. The intervention lasts 6 months followed by a 6-month step-down period.
  Interventions: Other: Replicating Effective Programs plus External Facilitation
- Educational Materials (Placebo Comparator): Dissemination of available materials explaining the Collaborative Chronic Care Model and implementation tools. Sites randomized to delay initiation of facilitation will have these materials plus technical assistance for 4 or 8 months prior to full implementation facilitation.
  Interventions: Other: Educational Materials

INTERVENTIONS:
Other: Replicating Effective Programs plus External Facilitation — Packaging, training and technical assistance according to the Replicating Effective Programs model plus External Facilitation
  Other Names: REP-F
  Arms: Implementation Facilitation
Other: Educational Materials — Dissemination of educational materials on the collaborative chronic care model for 4 or 8 months prior to cross-over to REP-F
  Arms: Educational Materials

SUMMARY:
This randomized program evaluation is undertaken in conjunction with the Department of Veterans Affairs (VA) Office of Mental Health Operations (OMHO) and the Quality Enhancement Research Initiative. It is designed to answer two related questions: (1) Can an evidence-based implementation strategy using the Center for Disease Control (CDC)'s Replicating Effective Programs plus External Facilitation (REP-F) enhance the adoption of team-based care in VA General Mental Health (GMH) Clinics, and (2) Does the establishment of such teams via implementation enhance Veterans' health status, satisfaction, and perceptions of care? The model for team-based care is the evidence-based Collaborative Chronic Care Model (CCM).

In conjunction with a nation-wide roll-out of the VA's Behavioral Health Interdisciplinary Program team (BHIP) initiative, the investigators have structured a randomized, controlled program evaluation to answer these questions. Specifically, using a stepped wedge design the investigators will randomize 9 VAMCs that have requested support in establishing a BHIP to 1 of 3 waves of REP-F support: immediate implementation support vs. 4-month vs. 8-month wait with dissemination of CCM materials (3 sites per wave). Fidelity and health outcome measures will be collected in a repeated measures design at 6-month intervals, and analyzed with general linear modeling.

DETAILED DESCRIPTION:
Based on an internal system-wide review of mental health services and the Mental Health Action Plan submitted to Congress in November, 2011, the Office of Mental Health Operations (OMHO) has undertaken an effort to establish behavioral health interdisciplinary plans (BHIPs), which are intended to provide General Mental Health (GMH) care throughout the Department of Veterans Affairs (VA). The BHIP goal is to build effective interdisciplinary teams, which will provide the majority of care for Veterans in GMH. It is now expected that every Veterans Affairs Medical Center (VAMC) establish at least one BHIP in the current initial phase (begun in late fiscal year 2013), and that the effort scale-up subsequently. Not surprisingly, progress has been uneven.

In 2015 OMHO incorporated the Collaborative Chronic Care Model (CCM) as an evidence-based model by which to structure BHIPs. Consistent with BHIP goals, CCMs were developed to provide anticipatory, continuous, collaborative, evidence-based care. CCMs consist of 6 elements: delivery system redesign, use of clinical information systems, provider decision support, patient self-management support, linkage to community resources, and healthcare organization support. Replicating Effective Programs with External Facilitation (REP-F) has been shown to be effective in implementing complex care models, including CCMs for mental health, both within and beyond VA.

Thus in conjunction with OMHO, the investigators propose this project with the Specific Aim of evaluating the impact of REP-F in implementing CCM-based BHIPs and their effect on Veteran health status. The investigators propose a Hybrid Type III implementation-effectiveness stepped wedge controlled trial, specifically hypothesizing that:

H1: REP-F-based implementation to establish CCM-based BHIPs, compared to existing centralized technical assistance will result in: (H1a) increased Veteran perceptions of CCM-based care, (H1b) higher rates of achieving national BHIP clinical fidelity measures (implementation outcomes), and (H1c) higher provider ratings of the presence of CCM elements.

H2: CCM-based BHIPs, supported by REP-F implementation, will result in improved Veteran health outcomes compared to BHIPs supported by dissemination material alone (intervention outcomes).

The investigators will utilize the national BHIP rollout as a vehicle for this project. Using a stepped wedge design the investigators will randomize 9 VAMCs that have requested support in establishing a BHIP to 1 of 3 waves of REP-F support: immediate implementation support vs. 4-month vs. 8-month wait with dissemination of CCM materials (3 sites per wave). Fidelity and health outcome measures will be collected in a repeated measures design at 6-month intervals, and analyzed with general linear modeling.

ELIGIBILITY:
Inclusion Criteria:

At least three visits to the General Mental Health Clinic's BHIP team in prior year

Exclusion Criteria:

Chart evidence of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1112 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Bauer, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woltmann E, Grogan-Kaylor A, Perron B, Georges H, Kilbourne AM, Bauer MS. Comparative effectiveness of collaborative chronic care models for mental health conditions across primary, specialty, and behavioral health care settings: systematic review and meta-analysis. Am J Psychiatry. 2012 Aug;169(8):790-804. doi: 10.1176/appi.ajp.2012.11111616. PMID 22772364
- [Background] Miller CJ, Grogan-Kaylor A, Perron BE, Kilbourne AM, Woltmann E, Bauer MS. Collaborative chronic care models for mental health conditions: cumulative meta-analysis and metaregression to guide future research and implementation. Med Care. 2013 Oct;51(10):922-30. doi: 10.1097/MLR.0b013e3182a3e4c4. PMID 23938600
- [Background] Waxmonsky J, Kilbourne AM, Goodrich DE, Nord KM, Lai Z, Laird C, Clogston J, Kim HM, Miller C, Bauer MS. Enhanced fidelity to treatment for bipolar disorder: results from a randomized controlled implementation trial. Psychiatr Serv. 2014 Jan 1;65(1):81-90. doi: 10.1176/appi.ps.201300039. PMID 24129806
- [Derived] Sullivan JL, Kim B, Miller CJ, Elwy AR, Drummond KL, Connolly SL, Riendeau RP, Bauer MS. Collaborative chronic care model implementation within outpatient behavioral health care teams: qualitative results from a multisite trial using implementation facilitation. Implement Sci Commun. 2021 Mar 24;2(1):33. doi: 10.1186/s43058-021-00133-w. PMID 33762023
- [Derived] Connolly SL, Sullivan JL, Ritchie MJ, Kim B, Miller CJ, Bauer MS. External facilitators' perceptions of internal facilitation skills during implementation of collaborative care for mental health teams: a qualitative analysis informed by the i-PARIHS framework. BMC Health Serv Res. 2020 Mar 4;20(1):165. doi: 10.1186/s12913-020-5011-3. PMID 32131824
- [Derived] Lew RA, Miller CJ, Kim B, Wu H, Stolzmann K, Bauer MS. A method to reduce imbalance for site-level randomized stepped wedge implementation trial designs. Implement Sci. 2019 May 3;14(1):46. doi: 10.1186/s13012-019-0893-3. PMID 31053157
- [Derived] Bauer MS, Miller CJ, Kim B, Lew R, Stolzmann K, Sullivan J, Riendeau R, Pitcock J, Williamson A, Connolly S, Elwy AR, Weaver K. Effectiveness of Implementing a Collaborative Chronic Care Model for Clinician Teams on Patient Outcomes and Health Status in Mental Health: A Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190230. doi: 10.1001/jamanetworkopen.2019.0230. PMID 30821830
- [Derived] Bauer MS, Miller C, Kim B, Lew R, Weaver K, Coldwell C, Henderson K, Holmes S, Seibert MN, Stolzmann K, Elwy AR, Kirchner J. Partnering with health system operations leadership to develop a controlled implementation trial. Implement Sci. 2016 Feb 24;11:22. doi: 10.1186/s13012-016-0385-7. PMID 26912342

RESULTS

PARTICIPANT FLOW:
Groups:
- Veteran Participants: In this stepped wedge design that is not a randomized control trial (RCT), those eligible BHIP team-treated veterans randomly selected for telephone interview for health status measures. Primary analyses were within-subject.
- Provider Participants: In this stepped wedge design that is not a randomized control trial (RCT), BHIP team clinicians who participated in team function survey. Primary analyses were within-subject.
Period: Overall Study
Arm/Group | Veteran Participants | Provider Participants
Started | 1050 (This is a quasi-experimental design, not a RCT. 1050 veterans did 1436 interviews at 3 time points.) | 62
0 Month Timepoint (t0) | 593 | 40
6 Month Timepoint (t6) | 66 (593 participants started at 0 months; 188 repeated and 66 participants added at 6 months timepoint.) | 0
12 Month Timepoint (t12) | 391 (91 continued from 0 months (t0), 16 from 6 months (t6), 91 from t0 & t6; 391 added at 12 months.) | 22 (22 new providers completed at 12 months; 21 completed at both 0 and 12 months. 19 completed only T0.)
Completed | 1050 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Most baseline demographic characteristics of provider participants not collected.
Groups:
- Veteran Participants: In this stepped wedge design, those eligible BHIP team-treated veterans randomly selected for telephone interview for health status measures. Primary analyses were within-subject.
- Provider Participants: In this stepped wedge design, BHIP team clinicians who participated in team function survey. Primary analyses were within-subject.
- Total: Total of all reporting groups
Arm/Group | Veteran Participants | Provider Participants | Total
Number analyzed (Participants) | 1050 | 62 | 1112
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.7) | 49.6 (9.9) | 52.405 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 35 | 245
  Male | 840 | 27 | 867
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Veteran participants self-reported as one or more races/ethnicities so total exceeds 1050. "Other" includes Alaska Native or Native American, Native Hawaiian or Pacific Islander, Asian, and Other. Minority groups all who reported one or more categories besides "White/Caucasian." Eligible Veterans data not self-reported, from VA Corporate Data Warehouse (CDW). Population: Provider ethnicity not collected.
  Participants
    White: number analyzed (Participants) | 1050 | 0 | 1050
    White | 825 |  | 825
    Black: number analyzed (Participants) | 1050 | 0 | 1050
    Black | 159 |  | 159
    Other: number analyzed (Participants) | 1050 | 0 | 1050
    Other | 26 |  | 26
    Hispanic or Latino: number analyzed (Participants) | 1050 | 0 | 1050
    Hispanic or Latino | 97 |  | 97
    Minority: number analyzed (Participants) | 1050 | 0 | 1050
    Minority | 275 |  | 275
Marital Status (currently married) [Count of Participants; unit: Participants] — Population: Marital status not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 487 |  | 487
Employment Status (full-time, part-time, or self- employed) [Count of Participants; unit: Participants] | 532 | 62 | 594
Rural residence (rural and highly rural) [Count of Participants; unit: Participants] — Population: Residence rurality not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 227 |  | 227
Period of service (Gulf War or later, 1990-present) [Count of Participants; unit: Participants] — Population: Military service not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 497 |  | 497
VA disability % (>= 50%) [Count of Participants; unit: Participants] — Population: VA disability percentage (amount of disability assigned to VA patients that determines amount of care financially covered by VA). Not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 844 |  | 844
Depression or anxiety disorder [Count of Participants; unit: Participants] — Population: Diagnoses not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 592 |  | 592
Serious Mental Illness (bipolar spectrum or schizophrenia) [Count of Participants; unit: Participants] — Population: Diagnoses not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 340 |  | 340
Post traumatic stress disorder [Count of Participants; unit: Participants] — Population: Diagnoses not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 474 |  | 474
Substance use disorder [Count of Participants; unit: Participants] — Population: Diagnoses not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 169 |  | 169
Number of active mental health diagnoses (mean + sd) [Mean (Standard Deviation); unit: diagnoses] — Population: Diagnoses not collected for providers.
  diagnoses
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 2.2 (1.4) |  | 2.2 (1.4)
Number of active medical diagnoses (mean + sd) [Mean (Standard Deviation); unit: diagnoses] — Population: Diagnoses not collected for providers.
  diagnoses
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 1.2 (1.3) |  | 1.2 (1.3)
Mental health hospitalization in prior year [Count of Participants; unit: Participants] — Population: Hospitalizations not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 36 |  | 36
Medical-surgical hospitalization in prior year [Count of Participants; unit: Participants] — Population: Hospitalizations not collected for providers.
  Participants
    number analyzed (Participants) | 1050 | 0 | 1050
    (all) | 73 |  | 73
Team Development Measure (TDM) [Mean (Standard Deviation); unit: scores on a scale] — Team Development Measure (TDM) is a survey assessing team function at baseline and during the second six months of implementation using the four subscales with items rated from strongly agree to strongly disagree: Communication, Cohesion, Role Clarity, and Team Primacy (prioritizing team over individual goals). The percentage of team members agreeing or strongly agreeing with each statement was calculated, then averaged across all statements for a mean percentage for each subscale. Range of percentage was 0-100. Missing: cohesion (3); communication (2); role clarity (1); team primacy (0). Population: Not collected for veterans participants (n=1050).
  scores on a scale
    Cohesion: number analyzed (Participants) | 0 | 59 | 59
    Cohesion |  | 84.0 (20.8) | 84.0 (20.8)
    Communication: number analyzed (Participants) | 0 | 60 | 60
    Communication |  | 83.3 (24.6) | 83.3 (24.6)
    Role Clarity: number analyzed (Participants) | 0 | 61 | 61
    Role Clarity |  | 53.4 (26.9) | 53.4 (26.9)
    Team Primacy: number analyzed (Participants) | 0 | 62 | 62
    Team Primacy |  | 50.0 (37.6) | 50.0 (37.6)

OUTCOME MEASURES:

1. Primary Outcome: Veterans RAND-12 Mental Component Score (VR-12 MCS)
Description: Veterans RAND-Mental Component Score: Overall self-rated mental health status over past two weeks among Veteran participants. Possible scores of minimum 0 and maximum 50. Higher is better. Administered with items for Veterans RAND-Physical Component Score.
Time Frame: one year
Population: Adjusted mixed model of single group with repeated event. Number Analyzed = number of participants with available data at the specified time points. 1050 participants completed 1436 interviews across one or more time points: t0, t6, t12. 589 started at t0 (missing=4); 65 added at t6 (missing=1); 386 added at t12 (missing=5).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veteran Participants
Number analyzed (Participants) | 1050
score on a scale
  Baseline (T0): number analyzed (Participants) | 589
  Baseline (T0) | 36.82 (14.78)
  Six Month Timepoint (T6): number analyzed (Participants) | 65
  Six Month Timepoint (T6) | 36.24 (14.26)
  Final Twelve Month Timepoint (T12): number analyzed (Participants) | 386
  Final Twelve Month Timepoint (T12) | 37.25 (14.07)
Statistical Analysis 1: Comparison: Veteran Participants; Test type: Superiority; p < 0.01, Mixed Models Analysis — Adjusted for multiple comparisons (Bonferroni four comparisons); Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.26 to 1.5]
Statistical Analysis 2: Comparison: Veteran Participants; Among Veteran participants,we used a linear contrast comparing a) those with complex clinical presentations, defined as receiving treatment for three or more mental health diagnoses in the prior year to b) those with two or fewer diagnoses during the facilitation year from T0 to T12; Test type: Superiority; p < 0.001, Regression, Linear — Adjusted for comparisons (Bonferroni for 4 comparisons.); Mean Difference (Final Values) = 5.03, 95% CI 2-sided [2.24 to 7.82]

2. Secondary Outcome: Veterans RAND-12 Physical Component Scores (VR-12 PCS)
Description: Veterans RAND-Physical Component Score: Overall self-rated physical health status over past two weeks among Veteran participants. Possible scores of minimum 0 and maximum 50. Higher is better. Administered with items for Veterans RAND-Mental Component Score.
Time Frame: One year
Population: Adjusted mixed model of a single group with repeated event. Number Analyzed = number of participants with available data and the specified time points. 1050 completed 1436 interviews across t0, t6, t12. 593 started at t0; 66 added at t6; 391 added at t12. None missing from survey. Site included as random effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veteran Participants
Number analyzed (Participants) | 1050
score on a scale
  T0: number analyzed (Participants) | 593
  T0 | 35.20 (13.11)
  T6: number analyzed (Participants) | 66
  T6 | 35.62 (12.61)
  T12: number analyzed (Participants) | 391
  T12 | 35.30 (12.31)
Statistical Analysis 1: Comparison: Veteran Participants; Test type: Superiority; p < 0.04, Mixed Models Analysis — Adjusted for comparison (Bonferroni for four comparisons.); Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.04 to 2.3]

3. Secondary Outcome: Satisfaction Index
Description: Satisfaction Index: Overall patient satisfaction with mental health services. Higher is better. Minimum score is 12, maximum score is 72.
Time Frame: One year
Population: Adjusted mixed model of a single group with repeated event. Number Analyzed = number of participants with available data and the specified time points. 1050 completed 1436 interviews across t0, t6, t12. 576 started at t0 (missing=17); 64 added at t6 (missing=2); 380 added at t12 (missing=11). Site included as random effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veteran Participants
Number analyzed (Participants) | 1050
score on a scale
  T0: number analyzed (Participants) | 576
  T0 | 52.94 (14.40)
  T6: number analyzed (Participants) | 64
  T6 | 53.26 (15.08)
  T12: number analyzed (Participants) | 380
  T12 | 52.78 (15.18)
Statistical Analysis 1: Comparison: Veteran Participants; Test type: Superiority; p > 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.2 to 0.9]

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: Recovery-oriented quality of life score. Higher is better. Minimum score 0, maximum score 100.
Time Frame: One year
Population: Adjusted mixed model of a single group with repeated event. Number Analyzed = number of participants with available data and the specified time points. 1050 completed 1436 interviews across t0, t6, t12. 577 started at t0 (missing=16), 63 added at t6 (missing=3); 380 added at t12 (missing=11). Site included as random effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veteran Participants
Number analyzed (Participants) | 1050
score on a scale
  Baseline (T0): number analyzed (Participants) | 577
  Baseline (T0) | 53.2 (19.33)
  Six Month Timepoint (T6): number analyzed (Participants) | 63
  Six Month Timepoint (T6) | 53.9 (20.82)
  Final Twelve Month Timepoint (T12): number analyzed (Participants) | 380
  Final Twelve Month Timepoint (T12) | 54.8 (19.65)
Statistical Analysis 1: Comparison: Veteran Participants; Test type: Superiority; p > 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.3 to 2.3]

5. Secondary Outcome: Patient Assessment of Chronic Illness Care (PACIC)
Description: Patient Assessment of Chronic Illness Care (PACIC): Veteran perception of coordination of and engagement with services. Higher is better. Minimum score is 1, maximum score is 33.
Time Frame: One year
Population: Adjusted mixed model of a single group with repeated event. Number Analyzed = number of participants with available data and the specified time points. 1050 completed 1436 interviews across t0, t6, t12. 582 started at t0 (missing=11); 65 added at t6 (missing=1); 384 added at t12 (missing=7). Site included as random effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veteran Participants
Number analyzed (Participants) | 1050
score on a scale
  T0: number analyzed (Participants) | 582
  T0 | 21.94 (6.35)
  T6: number analyzed (Participants) | 65
  T6 | 22.46 (6.57)
  T12: number analyzed (Participants) | 384
  T12 | 21.99 (6.40)
Statistical Analysis 1: Comparison: Veteran Participants; Test type: Superiority; p > 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.8]

6. Secondary Outcome: Team Development Measure (TDM)- Cohesion
Description: Mean percentage of participant provider team members who strongly agreed or agreed with the cohesion domain within the Team Development Measure.
  Measure Description: Team Development Measure (TDM) is a survey assessing team function at baseline and during the second six months of implementation using the four subscales with items rated from strongly agree to strongly disagree: Communication, Cohesion, Role Clarity, and Team Primacy (prioritizing team over individual goals). The percentage of team members agreeing or strongly agreeing with each statement was calculated, then averaged across all statements for a mean percentage for each subscale. Range of percentage was 0-100.
Time Frame: baseline and during stepdown (6-12 months)
Population: Total 62 mental health providers who completed survey. Number Analyzed = number of participants with available data at the specified time points for Cohesion domain (missing=3). 40 completed at 0 months (t0) and 43 completed at 12 months (t12). 21 new providers completed at t12; 22 completed at both t0 and t12. 19 completed only t0.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Participants
Number analyzed (Participants) | 59
score on a scale
  Baseline (T0): number analyzed (Participants) | 40
  Baseline (T0) | 84.0 (20.8)
  Follow-up/Final at Six to Twelve Months (T12): number analyzed (Participants) | 43
  Follow-up/Final at Six to Twelve Months (T12) | 84.5 (22.4)
Statistical Analysis 1: Comparison: Provider Participants; Test type: Superiority; p > 0.05, t-test, 2 sided; Paired; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.074 to 0.084]

7. Secondary Outcome: Team Development Measure (TDM)- Communication
Description: Mean percentage of participant team members who strongly agreed or agreed with the communication domain within the Team Development Measure.
  Measure Description: Measure Description: Team Development Measure (TDM) is a survey assessing team function at baseline and during the second six months of implementation using the four subscales with items rated from strongly agree to strongly disagree: Communication, Cohesion, Role Clarity, and Team Primacy (prioritizing team over individual goals). The percentage of team members agreeing or strongly agreeing with each statement was calculated, then averaged across all statements for a mean percentage for each subscale. Range of percentage was 0-100.
Time Frame: baseline and during stepdown (6-12 months)
Population: Total 62 mental health providers who completed survey. Number Analyzed = number of participants with available data and the specified time points for Communication domain (missing=2). 40 completed at 0 months (t0) and 43 completed at 12 months (t12). 21 new providers completed at t12; 22 completed at both t0 and t12. 19 completed only t0.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Participants
Number analyzed (Participants) | 60
score on a scale
  Baseline (T0): number analyzed (Participants) | 40
  Baseline (T0) | 83.3 (24.6)
  Follow-up/Final at Six to Twelve Months (T12): number analyzed (Participants) | 43
  Follow-up/Final at Six to Twelve Months (T12) | 84.4 (20.6)
Statistical Analysis 1: Comparison: Provider Participants; Test type: Superiority; p > 0.05, t-test, 2 sided; Paired; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.056 to 0.077], Standard Deviation 0.206

8. Secondary Outcome: Team Development Measure (TDM)- Role Clarity
Description: Mean percentage of participant team members who strongly agreed or agreed with the role clarity domain within the Team Development Measure.
  Measure Description: Team Development Measure (TDM) is a survey assessing team function at baseline and during the second six months of implementation using the four subscales with items rated from strongly agree to strongly disagree: Communication, Cohesion, Role Clarity, and Team Primacy (prioritizing team over individual goals). The percentage of team members agreeing or strongly agreeing with each statement was calculated, then averaged across all statements for a mean percentage for each subscale. Range of percentage was 0-100. Missing: cohesion (3); communication (2); role clarity (1); team primacy (0).
Time Frame: baseline and during stepdown (6-12 months)
Population: Total 62 mental health providers who completed survey.Number Analyzed = number of participants with available data and the specified time points for Role Clarity domain (missing= 1). 40 completed at 0 months (t0) and 43 completed at 12 months (t12). 21 new providers completed at t12; 22 completed at both t0 and t12. 19 completed only t0.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Participants
Number analyzed (Participants) | 61
score on a scale
  Baseline (T0): number analyzed (Participants) | 40
  Baseline (T0) | 53.4 (26.9)
  Follow-up/Final at Six to Twelve Months (T12): number analyzed (Participants) | 43
  Follow-up/Final at Six to Twelve Months (T12) | 68.7 (28.7)
Statistical Analysis 1: Comparison: Provider Participants; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired; Mean Difference (Final Values) = 0.153, 95% CI 2-sided [0.044 to 0.262]

9. Secondary Outcome: Team Development Measure (TDM)- Team Primacy
Description: Mean percentage of participant team members who strongly agreed or agreed with the team primacy domain within the Team Development Measure.
  Measure Description: Team Development Measure (TDM) is a survey assessing team function at baseline and during the second six months of implementation using the four subscales with items rated from strongly agree to strongly disagree: Communication, Cohesion, Role Clarity, and Team Primacy (prioritizing team over individual goals). The percentage of team members agreeing or strongly agreeing with each statement was calculated, then averaged across all statements for a mean percentage for each subscale. Range of percentage was 0-100. Missing: cohesion (3); communication (2); role clarity (1); team primacy (0).
Time Frame: baseline and during stepdown (6-12 months)
Population: Total 62 mental health providers who completed survey. Number Analyzed = number of participants with available data and the specified time points for Team Primacy (0 missing). 40 completed at 0 months (t0) and 43 completed at 12 months (t12). 21 new providers completed at t12; 22 completed at both t0 and t12. 19 completed only t0.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Participants
Number analyzed (Participants) | 62
score on a scale
  Baseline (T0): number analyzed (Participants) | 40
  Baseline (T0) | 50.0 (37.6)
  Follow-up/Final at Six to Twelve Months (T12): number analyzed (Participants) | 43
  Follow-up/Final at Six to Twelve Months (T12) | 68.6 (28.7)
Statistical Analysis 1: Comparison: Provider Participants; Test type: Superiority; p < 0.01, t-test, 2 sided; Paired; Mean Difference (Final Values) = 0.186, 95% CI 2-sided [0.083 to 0.289]

10. Secondary Outcome: Mental Health Hospitalization Rates
Description: Quarterly indicator (0 not hospitalized or 1 hospitalized) for mental health hospitalization in the prior three months.
Time Frame: Two years
Population: All eligible patients were coded for hospitalization yes/no in each quarter.
Measure: Least Squares Mean (95% Confidence Interval); unit: beta coefficient
Groups:
- Eligible Veterans: In this stepped wedge design, all eligible BHIP team-treated veterans were utilized for hospitalization rate analyses. Primary analyses were within-subject.
Arm/Group | Eligible Veterans
Number analyzed (Participants) | 1050
beta coefficient | -0.12 [-0.16 to -0.07]
Statistical Analysis 1: Comparison: Eligible Veterans; Test type: Superiority; p < 0.001, Mixed Models Analysis — Repeated patient binary outcome models for hospitalized (0/1) across 8 quarters; Adjusted (Bonferroni four comparisons); Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.16 to -0.07]

ADVERSE EVENTS:
Time Frame: Full duration of the study from March 2016 through April 2018, approximately 1 year and 1 month.
Groups:
- Veteran Participants: Veterans in quasi-experimental stepped wedge design.
- Provider Participants: Providers in mental health (MH) clinics who participated in survey.
Arm/Group | Veteran Participants | Provider Participants
All-Cause Mortality (participants affected / at risk) | 0/1050 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/1050 | 0/62
Other Adverse Events (participants affected / at risk) | 0/1050 | 0/62

LIMITATIONS AND CAVEATS:
All facilities received implementation support, randomized as to start time. There was thus no independent parallel control group. However, several validity checks were conducted to establish internal validity of positive findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT02543840/Prot_SAP_000.pdf